CLINICAL TRIAL: NCT00809302
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy and Safety of Three Doses of Aplindore MR (1, 3, and 6 mg Twice Daily) in Patients With Early Parkinson Disease (APLIED)
Brief Title: Efficacy and Safety Study of Aplindore in Patients With Early Parkinson Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Neurogen acquired by Ligand Pharmaceuticals - no further support for study. No safety concerns identified.
Sponsor: Neurogen Corporation (Industry)
Responsible Party: Ken Sprenger, MD, MBBCh, Vice President, Clinical Development and Operations, Neurogen Corporation
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Aplindore-211
Record Dates: First submitted 2008-12-15; First posted 2008-12-17 (Estimated); Last update posted 2009-08-28 (Estimated); Status verified 2009-08

CONDITIONS: Early Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): aplindore 2 mg MR total daily dose
  Interventions: Drug: aplindore MR tablets or Placebo
- 2 (Experimental): aplindore 6 mg MR total daily dose
  Interventions: Drug: aplindore MR tablets or Placebo
- 3 (Experimental): aplindore 12 mg MR total daily dose
  Interventions: Drug: aplindore MR tablets or Placebo
- 4 (Placebo Comparator): Placebo
  Interventions: Drug: aplindore MR tablets or Placebo

INTERVENTIONS:
Drug: aplindore MR tablets or Placebo — aplindore MR tablets administered BID for about 13 weeks

SUMMARY:
This is a clinical trial to be conducted at multiple Parkinson Study Group (PSG) sites in the USA. Patients with early Parkinson disease will be randomly allocated to one of 4 arms in the study. The 4 arms include 3 arms with different doses of aplindore MR tablets and 1 placebo arm. The study drug will be taken twice a day (BID). The study is blinded and neither subjects, nor the investigators, will know what treatment the subject is receiving. Investigational study drug will be adjusted to the assigned dosage and then maintained at that dosage for the balance of the 12 week follow-up period. The entire study will take about 13 weeks. The study will assess the safety and tolerability of aplindore and measure how effective aplindore is in improving movement and other effects of Parkinson disease.

DETAILED DESCRIPTION:
One hundred and sixty eight patients will be randomly assigned to one of four investigational treatment regimens in this outpatient study. For active treatment arms, study drug will be titrated to the assigned dosage and then maintained for up to a 12 week follow-up period before receiving tapered doses in advance of study completion. Dosing will take place over a total of about 13 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 30 years old;
* Initial diagnosis of idiopathic PD must be within 5 years;
* At least two of the following cardinal signs must be present: bradykinesia, resting tremor, and rigidity;
* PD progression must be Stage 1 to 2.5 (inclusive) according to the modified Hoehn and Yahr classification system;
* Have a score on the MoCA of at least 26;
* Have a score on the Beck Depression Inventory II (BDI II) of less than 15;
* Have a screening UPDRS (Part III) motor score of at least 10;
* In good general health as determined by a thorough medical history and physical examination (including vital signs), neurological examination, 12-lead ECG, and clinical chemistry laboratory tests;
* Females of childbearing potential must be using an acceptable method of contraception and have a negative serum pregnancy test at the screening and baseline visits. Acceptable methods of contraception are oral, intrauterine, implantable, injectable contraceptives, double barrier methods or condoms impregnated with spermicide. After screening, subjects using oral contraceptive methods of contraception must agree to add an additional method until 30 days after the last dose of study medication. Women on oral contraceptives or using cervical rings must have been using them for at least 1 month before the screening visit;
* Male subjects with partners of childbearing potential must use adequate contraception during the study and for 3 months after the study;
* Females receiving hormone replacement therapy must be on a stable regimen for at least 3 months;
* Able to read, understand, and provide written/dated informed consent before enrolling in the study, and must be willing to comply with all study procedures.

Exclusion Criteria:

* History or clinical features consistent with an atypical parkinsonian syndrome;
* History of surgical intervention for PD;
* History of severe allergic or anaphylactic reaction to any drug;
* History of allergies or known sensitivity, hypersensitivity, or severe adverse reaction (e.g., requiring abrupt discontinuation) to any drug similar to aplindore;
* Taking prescription drug therapy or over the counter medication for chronic medical conditions who have not been on stable doses for at least 1 month before the screening visit;
* Treated with L-dopa within 2 months before the baseline visit or who have had cumulative treatment exceeding 2 months;
* Have taken dopamine agonist therapy within 1 month before the baseline visit or who have taken dopamine agonist therapy for a cumulative period exceeding 2 months;
* Are receiving amantadine, anticholinergics, or monoamine oxidase B inhibitors who have not been taking stable doses for at least 2 months before the baseline visit;
* A clinically significantly abnormal clinical laboratory value as judged by the investigator or a value that is disapproved by the study Clinical Monitor;
* A decrease in either systolic blood pressure of at least 40 mmHg or a decrease in diastolic blood pressure of at least 20 mmHg following 5 minutes supine and 2 minutes standing, at or within 6 months before the baseline visit;
* Clinically significant ECG findings, including prolonged QTcF intervals (>450 msec for men, >470 msec for women);
* Evidence of clinically significant unstable allergic (except for untreated, asymptomatic, seasonal allergies at time of dosing), hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, or neurological disease;
* History of basal or squamous cell skin cancers or carcinoma in situ of the cervix within 2 years before the screening visit are excluded; for all other cancer diagnoses, subjects with a history within 5 years before the screening visit are excluded;
* Any condition that may significantly affect drug absorption;
* Pregnant or lactating females;
* History or evidence of drug abuse or alcoholism as defined by DSM-IV TR within 12 months before the baseline visit or evidence of current withdrawal from drugs or alcohol before the baseline visit;
* Prior exposure to aplindore;
* Received any investigational drug within 60 days before the baseline visit.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-12; Primary Completion 2009-08 (Estimated); Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline to end of treatment in the combined scores of Parts II and III of the UPDRS | 3 months

SECONDARY OUTCOMES:
The responder rate; Part II and Part III scores (separately) of the UPDRS; mean change from baseline in the modified Schwab and England Activities of Daily Living; time course in UPDRS and in modified S&E-ADL; safety and tolerability of aplindore MR | 3 months

CONTACTS AND LOCATIONS:
Locations (25):
- United States (25):
  - University of Alabama At Birmingham (052), Birmingham, Alabama
  - Mayo Clinic Arizona (060), Scottsdale, Arizona
  - The Parkinson's Institute (012), Sunnyvale, California
  - Colorado Neurological Institute (052), Englewood, Colorado
  - Associated Neurologists, PC (190), Danbury, Connecticut
  - Eastern Connecticut Neurology Specialists (215), Manchester, Connecticut
  - Institute for Neurodegenerative Disorders (034), New Haven, Connecticut
  - Parkinson's Disease & Movement Disorders Center of Boca Raton (196), Boca Raton, Florida
  - University of Miami (014), Miami, Florida
  - University of South Florida (019), Tampa, Florida
  - Southern Illinois University (138), Springfield, Illinois
  - University of Kentucky (172), Lexington, Kentucky
  - University of Louisville (087), Louisville, Kentucky
  - Ochsner Clinic Foundation (207), New Orleans, Louisiana
  - LSU Health Science Center Shreveport (132), Shreveport, Louisiana
  - Boston University (040), Boston, Massachusetts
  - Washington University (027), St Louis, Missouri
  - Albany Medical College (037), Albany, New York
  - University of Rochester (001), Rochester, New York
  - Duke University Medical Center (119), Durham, North Carolina
  - University of Cincinnati/Cincinnati Children's Hospital (089), Cincinnati, Ohio
  - University of Pennsylvania (018), Philadelphia, Pennsylvania
  - Baylor College of Medicine (007), Houston, Texas
  - Booth Gardner Parkinson's Care Center (220), Kirkland, Washington
  - Medical College of Wisconsin (104), Milwaukee, Wisconsin